CLINICAL TRIAL: NCT00336271
Title: The Effects of Coffee
Status: Completed | Type: Observational
Sponsor: American University (Other)
Other Study IDs: 010
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Healthy Subjects
Keywords: coffee; caffeine; healthy subjects

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
In this study, participants will be eligible to participate in a paid research study that will examine the effects of regular coffee drinking. The study takes approximately 2 hours total, 55 min. on 2 separate days. Participants will be asked to do computer tasks and drink only coffee provided to them during the study.

DETAILED DESCRIPTION:
The purpose of the experiment is to evaluate how coffee affects different individuals while completing computer tasks. If an individual agrees to participate, particpants will be asked to come to the laboratory to drink coffee on 2 days. During each visit, participants will be asked to drink coffee, complete forms, and perform computer tasks. To be eligible to participate, participants must be medically healthy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be regular coffee drinkers.

For more information or to set up an appointment, please send a contact number (and a convenient time to call) via e-mail and a BPHP laboratory member will contact you or call the BPHP laboratory at the number listed below.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-04; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Moore, B.S., Principal Investigator — American University; Laura Juliano, Ph.D., Study Director — American University
Locations (1):
- Room 137 Asbury Building-American University, Washington D.C., District of Columbia, United States